CLINICAL TRIAL: NCT00364871
Title: Phase 2, Multicenter, Randomized, Double Blind, Placebo Controlled Study of Combination Therapy for Safety and Efficacy in Subjects With Uncomplicated Obesity
Brief Title: Efficacy and Safety Study of Combination Therapy to Treat Uncomplicated Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Eduardo Dunayevich, MD, Orexigen Therapeutics, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NB201
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 (Experimental): Bupropion SR (400 mg/day) plus Naltrexone (48 mg/day)
  Interventions: Drug: naltrexone and bupropion SR
- 2 (Experimental): Bupropion SR (400 mg/day) plus Naltrexone (16 mg/day)
  Interventions: Drug: naltrexone and bupropion SR
- 3 (Active Comparator): Bupropion SR (400 mg/day)
  Interventions: Drug: naltrexone and bupropion SR
- 4 (Active Comparator): Naltrexone (48 mg/day)
  Interventions: Drug: naltrexone and bupropion SR
- 5 (Placebo Comparator): B-Placebo plus N-Placebo
  Interventions: Drug: naltrexone and bupropion SR
- 6 (Placebo Comparator): B-Placebo plus N-Placebo
  Interventions: Drug: naltrexone and bupropion SR
- 7 (Experimental): Bupropion SR (400 mg/day) plus Naltrexone (32 mg/day)
  Interventions: Drug: naltrexone and bupropion SR

INTERVENTIONS:
Drug: naltrexone and bupropion SR — naltrexone 16, 32 or 48 mg/day and bupropion SR 400 mg/day

SUMMARY:
The purpose of this study is to determine the efficacy and safety of 3 combinations of naltrexone and bupropion SR compared to naltrexone alone, bupropion SR alone or placebo.

DETAILED DESCRIPTION:
A completed proof of concept study, OT-101 (Data on File, Orexigen Therapeutics, 2005), demonstrated that a combination of 300 mg bupropion SR and 50 mg naltrexone was associated with greater weight loss than bupropion SR alone, naltrexone alone, or placebo in subjects with uncomplicated obesity.

The hypothesis for the current trial is that by adjusting the doses and titration schedules of bupropion SR and naltrexone greater efficacy and improved tolerability can be achieved. In this trial, a higher dose of bupropion and 2 lower doses of naltrexone than utilized in the previous trial (OT-101) will be evaluated. The doses of both drugs will be titrated over 4 weeks and administered twice a day. There are 2 cohorts. At each site, cohort 2 recruitment began as soon as cohort 1 enrollment was completed. Cohort 1 treatment groups are (60 per group):

* Group 1: Bupropion SR (400 mg/day) plus Naltrexone (48 mg/day)
* Group 2: Bupropion SR (400 mg/day) plus Naltrexone (16 mg/day)
* Group 3: Bupropion SR (400 mg/day) plus N-Placebo
* Group 4: B-placebo plus Naltrexone (48 mg/day)
* Group 5: B-Placebo plus N-Placebo

Cohort treatment 2 Groups are:

* Group 6: B-Placebo plus N-Placebo (n=20)
* Group 7: Bupropion SR (400 mg/day) plus Naltrexone (32 mg/day)(n=60)

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects, 18 to 60 years of age
* Have body mass index (BMI) of 30 to 40 kg/m2
* Free from clinically significant illness or disease as determined by medical history and physical examination
* Non-smoker and no use of tobacco or nicotine products for at least 6 months prior to baseline
* Normotensive (systolic <140 mm Hg; diastolic <90 mm Hg). Anti-hypertensive medications are allowed with the exception of adrenergic blockers, beta-blockers and clonidine. Medical regimen must be stable for at least 6 weeks
* LDL cholesterol < 190 mg/dL and triglycerides < 400 mg/dL. Medications for treatment of dyslipidemia are allowed as long as medical regimen has been stable for at least 6 weeks
* No clinically significant abnormality of serum albumin, blood urea nitrogen, creatinine, calcium and phosphorus
* Bilirubin, ALT and AST within 1.5 x ULN
* No clinically significant abnormality of hematocrit, white blood cell count, white cell differential, or platelets
* Fasting glucose less than 140 mg/dL on no hypoglycemic agents
* No clinically significant abnormality on urinalysis
* TSH within 1.5 x ULN, normal T3, if TSH below lower limit of normal
* Negative serum pregnancy test in women with intact uterus
* Score < 11 for depression and score < 11 for anxiety on Hospital Anxiety and Depression (HAD) Scale
* ECG: no clinically significant abnormality
* Score of zero on the Mood Assessment questionnaire and a response of "No" to the Bipolar Disorder Questions
* If female with child-bearing potential, must be non-lactating and agree to use effective contraception throughout the study period and 30 days after discontinuation of study drugs
* Able to comply with all required study procedures and schedule
* Willing and able to give written informed consent

Exclusion Criteria:

* Obesity of known endocrine origin (e.g., untreated hypothyroidism, Cushing's syndrome)
* Serious medical condition or medical condition that limits participation in the prescribed exercise program: (e.g. unstable cardiovascular disease including congestive heart failure, angina pectoris, and myocardial infarction; stroke; claudication; acute limb ischemia; acute renal or hepatic disorder; renal, hepatic or respiratory insufficiency)
* Active malignancy or history of malignancy (other than non-melanoma skin cancer or surgically cured cervical cancer) within 5 years of enrollment
* Serious psychiatric condition (e.g., any history of bipolar disorder, psychosis, suicidal attempt or post-partum depression; a history of major depression, suicidal ideation or antidepressant use within 1 year)
* Type I or Type II diabetes mellitus requiring pharmacotherapy
* Excluded concomitant medications: anorectic agents; weight loss agents; dietary supplements to promote muscle building, enhance mood, or reduce appetite; adrenergic blockers; beta blockers; anti-psychotic agents; clonidine; theophylline; cimetidine; oral corticosteroids; anti-depressant; topiramate; Depo-Provera®, smoking cessation agents; frequent, known use of opioid or opioid-like analgesics
* History of surgical intervention for obesity
* History of seizure disorder or predisposition to seizures (e.g., history of cerebrovascular accident, significant head trauma, brain surgery, skull fracture, subdural hematoma, or febrile seizures)
* History of bulimia or anorexia nervosa
* History of drug or alcohol abuse within 5 years
* History of treatment with bupropion, or naltrexone within 12 months
* History of hypersensitivity to bupropion, or naltrexone
* Use of drugs, herbs, or dietary supplements known to significantly affect body weight within one month of baseline
* Use of investigational drug, device or procedure within 90 days
* Participation in any previous clinical trial conducted by Orexigen Therapeutics
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 410 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percentage change in total body weight | baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (7):
- United States (7):
  - Scripps Clinic Del mar, San Diego, California
  - CSRA Partners in Health, Inc, Augusta, Georgia
  - UK Clinical Research Organization, Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Center for Nutrition and Preventive Medicine, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - MUSC Weight Management Center, Charleston, South Carolina